CLINICAL TRIAL: NCT01657539
Title: Effects of Yogurt Containing Bifidobacterium Animalis Ssp. Lactis dn- 1173010 Probiotics in the Composition of Biofilms and Saliva of Orthodontic Patients: a Crossover, Double-blind, Randomized and Placebo Controlled Clinical Trial.
Brief Title: Effect of Probiotics Containing Yogurts on the Composition of Biofilms in Patients Under Orthodontic Treatment
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Federal University of Pelotas (Other)
Collaborators: Pontificia Universidade Católica do Rio Grande do Sul (Other)
Responsible Party: Principal Investigator, Maximiliano Sergio Cenci, Coordinator of Clinical Trial, Graduate of Program of Dentistry, Federal University of Pelotas
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: UFPEL-PPGO0013
Record Dates: First submitted 2012-08-02; First posted 2012-08-06 (Estimated); Last update posted 2013-09-18 (Estimated); Status verified 2013-09

CONDITIONS: Dental Caries; Oral Health
MeSH Terms: conditions — Dental Caries | interventions — Yogurt; Probiotics

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (2):
- Probiotics (Experimental): Group of patients using yogurt containing probiotics during the experimental phase of the study.
  Interventions: Dietary Supplement: Yogurt containing probiotics
- Control Yogurt (Placebo Comparator): Group of patients that will use a placebo yogurt for providing comparison with the experimental group.
  Interventions: Dietary Supplement: Placebo yogurt

INTERVENTIONS:
Dietary Supplement: Yogurt containing probiotics — patients assigned to this group will use a yogurt containing Bifidobacterium animalis once a day during 14 days before evaluation of the outcomes.
  Other Names: yogurt containing Bifidobacterium animalis
  Arms: Probiotics
Dietary Supplement: Placebo yogurt — Patients will use a yogurt without probiotics once a day during 14 days before evaluation of outcomes
  Other Names: Yogurt without probiotics
  Arms: Control Yogurt

SUMMARY:
Aim: To assess in vivo if the intake of yogurt containing Bifidobacterium animalis ssp. lactis DN- 1173010 probiotic for a period of 2 weeks affects the salivary levels or biofilms of mutans streptococci and the lactobacilli of patients undergoing orthodontic treatment. Methods: A crossover, double-blind, randomized and placebo controlled clinical trial will be performed with 26 volunteers during 4 periods. During periods 2 and 4 (2 weeks each) the volunteers will have a daily ingestion of yogurt containing probiotic or of control yogurt which did not contain probiotic. Periods 1 and 3 were run-in and wash-out periods of 1 and 4 weeks, respectively. Experimental samples of saliva and biofilm will be collected from each participant at the end of each phase. Mutans streptococci, lactobacilli, total aciduric microorganisms, Candida spp. and total cultivable microorganisms will be counted. The values before and after the treatment will be compared with Wilcoxon's test (p<0.05).

ELIGIBILITY:
Inclusion Criteria:

* excellent oral health
* patients under bimaxillary orthodontic treatment

Exclusion Criteria:

* any chronic disease
* antibiotics and/or antimicrobial use in the previous 3 weeks
* topic fluoride or chlorhexidine use in the previous 3 weeks
* presence of cavitated or active carious lesions
* patients with intolerance to lactose.

Ages: 14 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2011-08; Primary Completion 2012-08 (Actual); Study Completion 2013-03 (Actual)

PRIMARY OUTCOMES:
Cariogenic bacteria reduction | 14 days
  The amount of cariogenic bacteria (mutans streptococci and lactobacilli) will be evaluated before and after the treatments for each patient

SECONDARY OUTCOMES:
Patient discomfort with the treatment | 14 days after intervention
  Patients were interviewed regarding any discomfort on the use of the treatments

CONTACTS AND LOCATIONS:
Overall Officials: Maximiliano S Cenci, PhD, Study Chair — Graduate Program in Dentistry, Federal University of Pelotas; Gabriela S Pinto, MSc, Principal Investigator — Graduate Program in Dentistry, Federal University of Pelotas
Locations (1):
- Graduate Program in Dentistry, Federal University of Pelotas, Pelotas, Rio Grande do Sul, Brazil